CLINICAL TRIAL: NCT01919242
Title: Postoperative Morbidity and Mortality After Gastrectomy for Gastric Cancer: Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0800
Record Dates: First submitted 2013-08-07; First posted 2013-08-08 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Patients Who Underwent Gastrectomy With Lymph Node Dissection for Gastric Cancer
MeSH Terms: interventions — Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- with morbidity: patients who suffered from any type of morbidity after surgery
  Interventions: Procedure: gastrectomy
- without morbidity: patients who did not suffer from any type of morbidity after surgery
  Interventions: Procedure: gastrectomy

INTERVENTIONS:
Procedure: gastrectomy — gastrectomy with D1 + lymph node dissection for clinically early gastric cancer, and gastrectomy with D2 lymph node dissection for clinically advanced gastric cancer

SUMMARY:
Gastric cancer is still one of the main health care issue and gastrectomy with lymph node dissection is the only chance to be cure. Even though the development and standardization of gastric cancer surgery, the morbidity of gastric cancer surgery was reported around 20% with less than 1% of mortality in East. In contrast, around 40% of morbidity and 10% of mortality was reported in West. There has been several indexes which can define the complications after surgery, but adapting it into clinical practice is sometimes difficult due to the heterogeneous opinion between surgeons. Thus for clear defining the complications after surgery, consensus between many surgeons and prospective cohort study is necessary. The purpose of this study is collecting the complications data after gastric cancer surgery and defining it with every week meeting by at least 6 or more surgeons' discussion.

ELIGIBILITY:
Inclusion Criteria:

* patients who had histologically confirmed gastric cancer and are going to underwent gastrectomy
* age over 20 years with agree to the study

Exclusion Criteria:

* withdrawal of their agreement
* vulnerable subjects (ex. pregnancy, disabled to decide by him or herself, cannot understand the study such as mental retardation or foreigner)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent gastrectomy with lymph node dissection for gastric cancer in Yonsei University Hospital, Seoul
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-01; Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
the type of complications and the incidence of it | within 30 days after operation, any case of re-admission
  the types of complication is classified into as follows: wound complications, intra-abdominal fluid collection or abscess, intra-luminal bleeding, intra-abdominal bleeding, intestinal obstruction, ileus, stricture of anastomosis, anastomosis leak, pancreatitis, pulmonary complications, urinary tract infection, renal dysfunction, hepatic dysfunction, cardiac dysfunction, endocrine dysfunction, miscellaneous complications. Each complication will be graded according to Clavian-Dindo classification. Re-admission or visiting emergency room will be checked and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University Health System, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Hartgrink HH, van de Velde CJ, Putter H, Bonenkamp JJ, Klein Kranenbarg E, Songun I, Welvaart K, van Krieken JH, Meijer S, Plukker JT, van Elk PJ, Obertop H, Gouma DJ, van Lanschot JJ, Taat CW, de Graaf PW, von Meyenfeldt MF, Tilanus H, Sasako M. Extended lymph node dissection for gastric cancer: who may benefit? Final results of the randomized Dutch gastric cancer group trial. J Clin Oncol. 2004 Jun 1;22(11):2069-77. doi: 10.1200/JCO.2004.08.026. Epub 2004 Apr 13. PMID 15082726
- [Background] Cuschieri A, Weeden S, Fielding J, Bancewicz J, Craven J, Joypaul V, Sydes M, Fayers P. Patient survival after D1 and D2 resections for gastric cancer: long-term results of the MRC randomized surgical trial. Surgical Co-operative Group. Br J Cancer. 1999 Mar;79(9-10):1522-30. doi: 10.1038/sj.bjc.6690243. PMID 10188901
- [Background] Wu CW, Hsiung CA, Lo SS, Hsieh MC, Chen JH, Li AF, Lui WY, Whang-Peng J. Nodal dissection for patients with gastric cancer: a randomised controlled trial. Lancet Oncol. 2006 Apr;7(4):309-15. doi: 10.1016/S1470-2045(06)70623-4. PMID 16574546
- [Background] Sasako M, Sano T, Yamamoto S, Kurokawa Y, Nashimoto A, Kurita A, Hiratsuka M, Tsujinaka T, Kinoshita T, Arai K, Yamamura Y, Okajima K; Japan Clinical Oncology Group. D2 lymphadenectomy alone or with para-aortic nodal dissection for gastric cancer. N Engl J Med. 2008 Jul 31;359(5):453-62. doi: 10.1056/NEJMoa0707035. PMID 18669424
- [Background] Bonenkamp JJ, Songun I, Hermans J, Sasako M, Welvaart K, Plukker JT, van Elk P, Obertop H, Gouma DJ, Taat CW, et al. Randomised comparison of morbidity after D1 and D2 dissection for gastric cancer in 996 Dutch patients. Lancet. 1995 Mar 25;345(8952):745-8. doi: 10.1016/s0140-6736(95)90637-1. PMID 7891484
- [Background] Cuschieri A, Fayers P, Fielding J, Craven J, Bancewicz J, Joypaul V, Cook P. Postoperative morbidity and mortality after D1 and D2 resections for gastric cancer: preliminary results of the MRC randomised controlled surgical trial. The Surgical Cooperative Group. Lancet. 1996 Apr 13;347(9007):995-9. doi: 10.1016/s0140-6736(96)90144-0. PMID 8606613
- [Background] Degiuli M, Sasako M, Ponti A, Soldati T, Danese F, Calvo F. Morbidity and mortality after D2 gastrectomy for gastric cancer: results of the Italian Gastric Cancer Study Group prospective multicenter surgical study. J Clin Oncol. 1998 Apr;16(4):1490-3. doi: 10.1200/JCO.1998.16.4.1490. PMID 9552056
- [Background] Kodera Y, Sasako M, Yamamoto S, Sano T, Nashimoto A, Kurita A; Gastric Cancer Surgery Study Group of Japan Clinical Oncology Group. Identification of risk factors for the development of complications following extended and superextended lymphadenectomies for gastric cancer. Br J Surg. 2005 Sep;92(9):1103-9. doi: 10.1002/bjs.4979. PMID 16106493
- [Background] Park DJ, Lee HJ, Kim HH, Yang HK, Lee KU, Choe KJ. Predictors of operative morbidity and mortality in gastric cancer surgery. Br J Surg. 2005 Sep;92(9):1099-102. doi: 10.1002/bjs.4952. PMID 15931657
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Strasberg SM, Linehan DC, Hawkins WG. The accordion severity grading system of surgical complications. Ann Surg. 2009 Aug;250(2):177-86. doi: 10.1097/SLA.0b013e3181afde41. PMID 19638919